CLINICAL TRIAL: NCT06266884
Title: The Effect of Kangaroo Care Training Given to Expectant Fathers in the Antenatal Period on Postpartum Father-Baby Attachment: Randomized Controlled Study
Brief Title: The Effect of Kangaroo Care on Father-Baby Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Emine Serap ÇAĞAN, Principal Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AgriIbrahimCecen
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Kangaroo Care; Attachment
Keywords: kangaroo care; Father-infant attachment
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: The contact numbers of the prospective fathers will be taken and a training video and presentation on kangaroo care will be sent via WhatsApp. Kangaroo care will be applied to the fathers in the experimental group during birth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo care group (Experimental): The contact numbers of the prospective fathers will be taken and a training video and presentation on kangaroo care will be sent via WhatsApp. Kangaroo care will be applied to the fathers in the experimental group during birth.
  Interventions: Other: Kangaroo care
- Control Group (No Intervention): After the fathers are informed that the birth has started, the postpartum questions prepared for the control group will be sent via WhatsApp and filled in by the fathers within the first 24 hours after birth. No other application will be applied to the control group. Father-Baby Attachment Scale questions will be sent to fathers via WhatsApp in the first and fourth months after birth and their answers will be received.

INTERVENTIONS:
Other: Kangaroo care — Kangaroo care is a safe and effective method in which the baby is placed in an upright position on the parent's bare chest, wearing only a diaper and a hat, and the baby's needs for nutrition, warmth, love and trust are met and provides positive interaction between the parent and the baby.
  Arms: Kangaroo care group

SUMMARY:
The aim of the research is to evaluate the attachment level of fathers who received kangaroo care training in the antenatal period and applied kangaroo care in the postpartum period to their babies in the first and fourth months.The research will be conducted in a randomized controlled experimental type with educational intervention. The research will be conducted at Islahiye State Hospital with 25 experimental and 25 control group fathers who meet the inclusion criteria. Fathers in the experimental group will be given kangaroo care training during the antenatal period and postpartum kangaroo care will be applied. No intervention will be made to the control group fathers. The Paternal-Infant Attachment Questionnaire (PPAQ) will be applied to fathers in both groups in the first and fourth months and the results will be compared.

DETAILED DESCRIPTION:
The aim of the research is to evaluate the attachment level of fathers who received kangaroo care training in the antenatal period and applied kangaroo care in the postpartum period to their babies in the first and fourth months.The research will be conducted in a randomized controlled experimental type with educational intervention. The research will be conducted at Islahiye State Hospital with 25 experimental and 25 control group fathers who meet the inclusion criteria. Fathers in the experimental group will be given kangaroo care training during the antenatal period and postpartum kangaroo care will be applied. No intervention will be made to the control group fathers. The Paternal-Infant Attachment Questionnaire (PPAQ) will be applied to fathers in both groups in the first and fourth months and the results will be compared.In the study, data will be collected using the father information form, postpartum questionnaire, postpartum kangaroo care competency checklist, kangaroo care application follow-up chart and father-baby attachment scale.

ELIGIBILITY:
Inclusion Criteria:

* 36-38. Coming to the hospital with her partner between weeks of gestation,
* Not having any physical and/or mental health problems,
* Not having a contagious disease transmitted by contact,
* Agreeing to participate in the research,
* Knowing Turkish and/or not having communication problems,
* Using Whatsapp application,
* Expecting a single baby

Exclusion Criteria:

* Being a foreign national, an immigrant or having communication problems,
* Having any physical and/or mental health problems,Having a transient contagious disease through contact,
* Refusing to participate in the research,
* Not using a phone and/or WhatsApp application,
* Expecting more than one baby

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Fathers will be included in the study.
Enrollment: 50 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Fathers' Attachment Level | from birth to 4 month after birth
  Father-infant attachment scale

CONTACTS AND LOCATIONS:
Locations (1):
- Agri Ibrahim Cecen University, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No